CLINICAL TRIAL: NCT02827903
Title: A Multi-center, Randomized, Double-blind, Phase III Clinical Trial to Compare the Efficacy and Safety of Metformin/Rosuvastatin Combination Therapy With Metformin or Rosuvastatin Monotherapy in Patients With Type 2 Diabetes and Dyslipidemia
Brief Title: Metformin/Rosuvastatin Combination Therapy With in Patients With Type 2 Diabetes and Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JLP-1310-P3-15
Record Dates: First submitted 2016-06-23; First posted 2016-07-11 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes; Dyslipidemia
Keywords: Metformin; Rosuvastatin; type 2 diabetes; dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Metformin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I (Experimental): Metformin + Rosuvastatin, Dosing to Type II DM with Dyslipidemia
  Interventions: Drug: Metformin + Rosuvastatin
- Group II (Active Comparator): Metformin + placebo, Dosing to Type II DM with Dyslipidemia
  Interventions: Drug: Metformin + placebo
- Group III (Active Comparator): Placebo + Rosuvastatin, Dosing to Type II DM with Dyslipidemia
  Interventions: Drug: placebo + Rosuvastatin

INTERVENTIONS:
Drug: Metformin + Rosuvastatin — Group I: Metformin + Rosuvastatin,
  Arms: Group I
Drug: Metformin + placebo — Group II: Metformin + placebo,
  Arms: Group II
Drug: placebo + Rosuvastatin — Group III: placebo + Rosuvastatin
  Arms: Group III

SUMMARY:
Compare the Efficacy and Safety of Metformin/Rosuvastatin Combination Therapy With Metformin or Rosuvastatin Monotherapy in Patients With Type 2 Diabetes and Dyslipidemia

DETAILED DESCRIPTION:
Multi-center, Randomized, Double-blind, Phase III clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years
* Type II DM with Dyslipidemia
* 6.5% ≤ HbA1c < 11%
* Triglyceride < 350mg/dL
* 100mg/dL ≤ LDL-C ≤ 250mg/dL
* FPG ≤ 270mg/dL

Exclusion Criteria:

* Type I DM
* Unstable angina, MI, Stroke, CABG with 6 month from screening
* SBP ≥ 180mmHg, DBP ≥ 110mmHg
* TSH > UNL
* Heart failure (NYHA class III/IV)
* Serum Creatinine > UNL or CLCr < 60 mL/min
* CK ≥ 2x UNL
* HIV positive
* BMI > 40 kg/m^2

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
LDL-C (% change) | 16 weeks from baseline
change of HbA1c | 16 weeks from baseline

CONTACTS AND LOCATIONS:
Locations (33):
- South Korea (33):
  - Buchoen St. mary's Hospital, Bucheon-si
  - SeJong Hostpital, Bucheon-si
  - SoonChunHyang University Bucheon Hospital, Bucheon-si
  - InJe University Busan paik Hospital, Busan
  - Inje University Haeundae paik hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Youngnam University Hostpital, Daegu
  - Daeheon Eulji Medical Center, Daejeon
  - KonYang University Hostpital, Daejeon
  - Chosun University Hospital, Gwangju
  - BunDang Jesang Hospital(DMC), Gyeonggi-do
  - Hallym University Sacred Heart hospital, Gyeonggi-do
  - HanYang University Guri Hospital, Gyeonggi-do
  - Inje University Ilsan paik hospital, Gyeonggi-do
  - Myoung Ji Hospital, Gyeonggi-do
  - Gachon Gil Hospital, Incheon
  - Inchoen St. mary's Hospital, Incheon
  - Eulji Hospital Nowon, Seoul
  - Hallym University Kangnam Sacred Heart hospital, Seoul
  - KangBuk SamSung Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - KonKuk University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - KyungHee University Hospital at Gangdong, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital(Famlily medicine), Seoul
  - Seoul National University Hospital, Seoul
  - Severance hospital, Seoul
  - SoonChunHayng University Hospital Seoul, Seoul
  - The catholic University of Korea YEOUIDO St mary's Hospital, Seoul
  - Korea University Guro hospital, Soeul
  - Ajou University hospital, Suwon
  - Wonju Severance Christian hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No